CLINICAL TRIAL: NCT00100828
Title: Phase II Trial of Irinotecan for Treatment of Metastatic Medullary Thyroid Cancer
Brief Title: Irinotecan in Treating Patients With Metastatic or Inoperable Thyroid Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to early stopping rule
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0459; P50CA096784 (NIH); P30CA006973 (NIH); JHOC-J0459; JHOC-04080402; CDR0000409567 (Other: other); 04-08-04-02 (Other: JHM IRB)
Record Dates: First submitted 2005-01-06; First posted 2005-01-07 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Head and Neck Cancer
Keywords: thyroid gland medullary carcinoma; recurrent thyroid cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Medullary; Thyroid Neoplasms | interventions — Irinotecan

ARMS (1):
- Irinotecan (Experimental)
  Interventions: Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well irinotecan works in treating patients with metastatic or inoperable thyroid cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with metastatic or inoperable locoregional medullary thyroid cancer treated with irinotecan.

Secondary

* Determine the safety and tolerability of this drug in these patients.

OUTLINE: Patients receive irinotecan IV on days 1 and 8. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Response is assessed after completion of 4 courses. Patients achieving complete response (CR) or partial response (PR) receive 2 additional courses beyond CR or PR. Patients who have stable disease receive up to 12 total courses.

PROJECTED ACCRUAL: A total of 33 patients will be accrued for this study.

ELIGIBILITY:
Inclusion

* Histologically confirmed medullary thyroid cancer
* Metastatic or inoperable locoregional disease
* Measurable disease by CT scan
* 18 years and over
* ECOG PS 0-1

Adequate lab functions including:

* Granulocyte count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Bilirubin < 1.5 mg/dL
* ALT and AST < 2.5 times upper limit of normal
* No unstable or uncompensated hepatic disease
* Creatinine clearance > 60 mL/min
* No unstable or uncompensated renal disease
* Negative pregnancy test
* More than 3 months since prior biologic therapy
* More than 3 months since prior chemotherapy
* No prior radiotherapy to > 25% of bone marrow
* More than 3 months since prior radiotherapy
* Recovered from prior oncologic or other major surgery
* More than 30 days since prior non-approved or investigational drugs

Exclusion:

* Patients with elevated calcitonin levels as the only measurement of disease are not eligible
* Unstable or uncompensated cardiovascular disease
* Unstable or uncompensated respiratory disease
* Pregnant or nursing
* Diarrhea ≥ grade 2 (antidiarrheals allowed)
* Other severe or uncontrolled systemic disease
* Other malignancy within the past 5 years except squamous cell or basal cell skin cancer or cervical cancer
* Illness that would preclude study participation
* Significant clinical disorder or laboratory finding that would preclude study participation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2004-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arlene A. Forastiere, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Groups:
- Irinotecan: irinotecan hydrochloride
Period: Overall Study
Arm/Group | Irinotecan
Started | 6
Completed (Trial closed due to early stopping rule and low enrollment.) | 0
Not Completed | 6
Not completed — Physician Decision | 6

BASELINE CHARACTERISTICS:
Arm/Group | Irinotecan
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (10.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: To determine the response rate of this regimen of irinotecan in patients with metastatic MTC
Time Frame: Every 2 cycles
Population: Study was closed to enrollment due to low accrual. Data was not collected for this outcome measure.
Arm/Group | Irinotecan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Irinotecan
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes